CLINICAL TRIAL: NCT02649244
Title: The Family Caregiver Training Program for Caregivers of People With Dementia: A Randomized Control Trial
Brief Title: The Family Caregiver Training Program for Caregivers of People With Dementia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Rosanne DiZazzo-Miller, PhD Candidate, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12181423Exp
Record Dates: First submitted 2016-01-04; First posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- The Family Caregiver Training Program (Experimental): The experimental group received a 2 hour intervention training on activities of daily throughout the early, middle, and late stages of dementia including communication, eating/feeding, nutrition, bathing, grooming, dressing, toileting, and transferring.
  Interventions: Behavioral: The Family Caregiver Training Program
- Standard Care (No Intervention): The control group received a 1 1/2 hour training, however the information was based on what has been deemed standard care by the Alzheimer's Association.

INTERVENTIONS:
Behavioral: The Family Caregiver Training Program — The intervention consisted of a two-hour PowerPoint® presentation throughout three modules (i.e., communication, eating/feeding, and nutrition; transferring and toileting; and dressing, bathing, and grooming). Each module was followed by a hands-on demonstration and practice session, including how to properly position and feed an adult, transfer from a seated position to another seated position, and a case study on modifications and assistance to provide during dressing and grooming.
  Arms: The Family Caregiver Training Program

SUMMARY:
The purpose of this study is to examine the effectiveness of the Family Caregiver Training Program for caregivers of people with dementia, using a pretest posttest randomized control trial with 3-month follow-up. The Family Caregiver Training Program will consist of 3-hours and hence, three modules over the course of one day. Module one will present information on communication, eating, and nutrition, module two will focus on transfers and toileting, and module three will focus on bathing, grooming, and dressing. The control group will receive standard care as relevant to dementia family caregivers including general information on the progression of dementia, and helpful resources as suggested by the Alzheimer's Association. A convenience sample of 36 family caregivers will be recruited by flyers posted throughout local area community boards and Alzheimer's Association media outlets. A repeated measures ANOVA will be used to assess the group differences in knowledge and confidence at three time points (pre-intervention, post-intervention, and 3-months post-intervention). Changes in caregiver burden, depression, quality of life, and occupational performance and satisfaction will be assessed 3-months post-intervention.

DETAILED DESCRIPTION:
The main research question asks to what extent does participation in a structured 3-hour training module (i.e., The Family Caregiver Training Program) focused on assisting family caregiver's with the ADLs of people with dementia effect caregiver knowledge and confidence, which in turn may effect caregiver burden, depression, quality of life, and occupational performance and satisfaction. Aim 1 will examine the relationship between the Family Caregiver Training Program intervention and knowledge of and confidence in the occupation of caregiving. Aim 2 will explore the relationship between the occupation of caregiving and person characteristics including burden, depression, and quality of life. Aim 3 will explore the relationship between the changes in the occupation of caregiving and changes in occupational performance.

A feasibility of the Family Caregiver Training Program was established using a single pre- post- test design. A significant improvement in caregiver knowledge was found in all three areas of training: communication/nutrition (N=53, p<0.001), transfers and toileting (N=46, p=0.003), and bathing and dressing (N=45, p=0.10) (DiZazzo-Miller, Samuel, Barnas, & Welker, 2014). This proposed study is built on the feasibility study, with the addition of confidence, burden, depression, quality of life, and occupational performance and satisfaction as outcomes using a random assignment to control group design.

A convenience sample of 36 family caregivers was recruited through flyers, newsletters, and Alzheimer's Association media outlets. The intervention group received one two-hour training that included three modules. Module one presented information on communication, eating/feeding and nutrition; module two focused on transfers and toileting; and module three focused on bathing, grooming, and dressing. The control group received standard care based upon a packet developed by the Alzheimer's Association for physicians to distribute to families and caregivers after receiving a diagnosis of dementia.

Results from this study will be generalizable to Metro-Detroit area family caregivers. Findings may offer information to enhance the caregiver training literature in the field of occupational therapy on the impact a community-based activity of daily living training can have with dementia family caregivers.

ELIGIBILITY:
Inclusion Criteria:

1. Primary family caregiver as providing at least 4 hours/day of care at least 5 days/week
2. At least 18 years of age
3. Able to read and understand the English language
4. Care recipients must have received an Alzheimer's or related dementia diagnosis

Exclusion Criteria:

1. Caregivers who provide less than 4 hours/day of care at least 5 days/week
2. Under 18 years of age
3. Unable to read or understand the English language
4. Have care recipients who have not received an Alzheimer's or related dementia diagnosis
5. Formally trained/paid caregivers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Caregiver Change in Activities of Daily Living Knowledge | Pretest (i.e., immediately before training) to Posttest (i.e., immediately after training-on the same day) and 3-Months Posttest.
  The ADL Knowledge Test is an 18-item, multiple-choice measure of caregiver assistance.
Caregiver Change in Confidence | Pretest (i.e., immediately before training) to Posttest (i.e., immediately after training-on the same day) and 3-Months Posttest.
  The Caregiver Confidence Scale (Lewis et al., 2010) is a modified nine-item confidence scale used to assess caregiver confidence in their skills for caring, understanding of the stages of dementia, and communication with their care recipient.

SECONDARY OUTCOMES:
The Zarit Burden Interview (22-item) | Pretest and 3-months posttest
  The Zarit Burden Interview (Zarit et al., 1980) is a measure of perceived caregiver burden.
The Beck Depression Inventory II | Pretest and 3-months posttest
  The Beck Depression Inventory-II (Beck, Steer, Ball, & Ranieri, 1996; Gallagher, Nies, & Thompson, 1982) was used to measure caregiver depression.
WHOQOL-BREF | Pretest and 3-months posttest
  The World Health Organization Quality of Life (Brief) measure (WHO-QOL-BREF) was used to measure four domains, including physical health, psychological, social relationships, and environment.
Occupational Performance | Pretest and 3-months posttest
  This scale consists of asking one question related to performance for each of the three ADL modules within the Family Caregiver Training Program using a Likert scale of 1 to 10 (1 as not at all and 10 as extremely) on how well caregivers perform their occupation of caregiving. This was adapted from the Canadian Occupational Performance Measure (COPM).
Occupational Satisfaction | Pretest and 3-months posttest
  This scale consists of asking one question related to satisfaction for each of the three ADL modules within the Family Caregiver Training Program using a Likert scale of 1 to 10 (1 as not at all and 10 as extremely) on how satisfied caregivers are with their occupation of caregiving. This was adapted from the Canadian Occupational Performance Measure (COPM).

REFERENCES:
- [Background] DiZazzo-Miller R, Samuel PS, Barnas JM, Welker KM. Addressing everyday challenges: feasibility of a family caregiver training program for people with dementia. Am J Occup Ther. 2014 Mar-Apr;68(2):212-20. doi: 10.5014/ajot.2014.009829. PMID 24581408